CLINICAL TRIAL: NCT06989580
Title: Clinical Data Collection to Develop Improved Arrhythmia and Heart Failure Management Using BIOMONITOR
Brief Title: BIO|CONCEPT.BIOMONITOR-HF Collect Clinical Data From Heart Failure Patients Using BIOMONITOR Devices With a Study Specific Research Software
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: HS068
Record Dates: First submitted 2025-04-17; First posted 2025-05-25 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Arrhythmia; Decompensated Heart Failure; Atrial Fibrillation
Keywords: Worsening Heart Failure (WHF)
MeSH Terms: conditions — Heart Failure; Arrhythmias, Cardiac; Atrial Fibrillation

STUDY DESIGN:
Intervention Model Description: Data collection
Masking Description: Only commercial features of the BIOMONITOR IV are open label. The additional sensor data recorded by the study software are blinded to investigators and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Other): All study participants receive the investigational device
  Interventions: Device: BIOMONITOR IV with study software

INTERVENTIONS:
Device: BIOMONITOR IV with study software — Participants are inserted with a BIOMONITOR IV which is then turned into the investigational device by replacing the firmware with the study software.

SUMMARY:
[Plain language]: Heart failure (HF) patients often experience irregular heartbeats, known as arrhythmias. Atrial fibrillation (AF) is common among HF patients and can worsen their condition, leading to strokes and higher death rates. Most of what we know about arrhythmias in HF comes from patients with devices like ICDs or CRTs, which help manage heart rhythms. However, this study focuses on HF patients who don't qualify for these devices.

Researchers use the BIOMONITOR IV, a device that tracks heart activity remotely over a long period. The goal is to understand how often arrhythmias occur in these patients and to develop a predictive algorithm for worsening HF (WHF). This algorithm could help doctors intervene early and improve treatment, reducing hospital visits and deaths related to WHF.

To make the BIOMONITOR IV more effective for HF management, its firmware is updated to collect additional data, such as fluid levels, breathing rate, and body position. These factors may be important for predicting WHF events.

DETAILED DESCRIPTION:
This study aims to collect clinical data with regard to the two main study objectives:

- Objective arrhythmia: Assess the incidence of arrhythmias and the contribution of the BIOMONITOR to arrhythmia diagnosis and subsequent treatment.

- Objective heart failure events: Collect data from BIOMONITOR sensors and relate them to the heart failure status for development of a predictive algorithm for worsening HF.

ELIGIBILITY:
Inclusion Criteria:

* Patient has diagnosed heart failure for ≥90 days and current symptoms compatible with NYHA class II-III (according to most recent assessment)
* At least ONE of the following:

At least one documented admission with a primary diagnosis of worsening heart failure within last 12 months prior to enrollment;

OR Unscheduled outpatient visit with increase of oral loop diuretics (more than 2-fold) or IV diuretic or ultrafiltration therapy for acute WHF within last 6 months prior to enrollment;

OR elevated NT-proBNP/BNP values within last 3 months prior to enrollment i.e.:

If LVEF >50% --> Patients in SR: >450 / >150 pg/ml; Patients with AF present: >900 / >300 pg/ml

If LVEF <50% --> Patients in SR: >900 / >300 pg/ml; Patients with AF present: >1800 / >450 pg/ml

* Ability to understand the nature of the study
* Willingness to provide written informed consent
* Ability and willingness to perform follow-up visits at the study site and via phone
* Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring concept

Exclusion Criteria:

* Implanted with pacemaker, ICD or CRT device or ICM
* Class I indication for a pacemaker, ICD or CRT according to current guidelines.
* Permanent or long-standing persistent AF
* Stroke, MI or PCI/CABG within 3 months prior to enrollment
* Patient is on chronic renal or peritoneal dialysis
* Patient has complex adult congenital heart disease
* Patient has active cancer involving chemotherapy, immunotherapy or radiation therapy
* Patient life expectancy is less than 1 year
* Age <18 years
* Patient is participating in any other device or drug trial that may interfere with the treatment or protocol of this study or may significantly affect the study outcomes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-08-22 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Heart failure events confirmed by WHF Adjudication Committee | Whole study conduct (approx. 3.5 years)
  * Heart failure hospitalization
  * Worsening heart failure event without hospitalization
Arrhythmias and subsequent therapeutic interventions | Whole study conduct (approx. 3.5 years)
  * Incidence of new diagnoses of arrhythmias, by type and therapeutic consequences
  * Percentage of patients for which the BIOMONITOR contributed to newly diagnosed arrhythmias
  * Percentage of patients for which the BIOMONITOR contributed to the decision to initiate an arrhythmia therapy

CONTACTS AND LOCATIONS:
Overall Officials: Thorsten Lewalter, Prof. Dr., Principal Investigator — Biotronik SE & Co. KG
Locations (2):
- Ziekenhuis Oost Limburg AV, Genk, Belgium
- Peter Osypka Herzzentrum, Munich, Germany

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data may be shared with qualified healthcare practitioners or academic researchers upon request and with permission of BIOTRONIK. Requests shall be sent to the Clinical Research Department of BIOTRONIK.
Time Frame: To be specified
Access Criteria: See above